CLINICAL TRIAL: NCT02631967
Title: A New Anastomotic Technique After Ileocecal Resection for Crohn's Disease. Kono-s Anastomosis vs Stapled Side-to-side Anastomosis: a Randomized Controlled Trial
Brief Title: Surgical Prevention of Anastomotic Recurrence by Excluding Mesentery in Crohn's Disease
Acronym: SuPREMeCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Luigi Bucci, Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211/15
Record Dates: First submitted 2015-11-29; First posted 2015-12-16 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Crohn Disease
Keywords: Crohn disease; ileocecal resection; anastomosis; Kono
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kono anastomosis (Experimental): Patients receiving Kono anastomosis
  Interventions: Procedure: Kono anastomosis
- Stapled side-to-side anastomosis (Experimental): Patients receiving stapled side-to-side anastomosis
  Interventions: Procedure: Stapled side-to-side anastomosis

INTERVENTIONS:
Procedure: Kono anastomosis — Kono anastomosis
  Arms: Kono anastomosis
Procedure: Stapled side-to-side anastomosis — Stapled side-to-side anastomosis
  Arms: Stapled side-to-side anastomosis

SUMMARY:
Kono and collegues have described a new anastomotic technique to restore bowel contintuity after ileocecal resection for Crohn's disease (CD).

This tecnique implies a hand-sewn ileocolic anastomosis, that involves exclusively the antimesenteric side of the bowel and that functionally acts as an end-to-end anastomosis.

In a retrospective study, the authors have shown that this anastomotic tecnique, when compared to stapled side-to-side anastomosis, significantly reduces the severity of endoscopic recurrence at 1 year after surgery and the rate of reoperation for anastomotic recurrence at 5 years after surgery.

Aim of this trial is to compare the outcomes of the Kono anastomosis with the ones achieved by the stapled side-to-side anastomosis, within a prospective randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease requiring ileocecal resection

Exclusion Criteria:

* age > 75 years
* age < 18 years
* inability to give the consent to the participation in the trial
* refusal to participate in the trial after receiving accurate information

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Grade of endoscopic recurrence | 6 Months
  Severity of endoscopic recurrence (graded according to Rutgeerts' score) at the site of anastomosis at 6 months after surgery.
Surgical recurrence | Up to 5 years
  Rate of patients requiring resection for anastomotic recurrence within 5 years after surgery

SECONDARY OUTCOMES:
Endoscopic recurrence | 6 months up to 5 years
  Presence of endoscopic recurrence
Grade of endoscopic recurrence | 6 months up to 5 years
  Severity of endoscopic recurrence at the site of anastomosis
Clinical recurrence | Up to 5 years
  Presence of clinical recurrence (according to Crohn's disease activity index)
Operating time | Intraoperatively
  Duration of the operation (min)
Anastomosis time | Intraoperatively
  Time (min) required to perform the anastomosis
Anastomotic leak | Up to 30 days
  Incidence of anastomotic leak
Surgical re-intervention | Up to 30 days
  Rate of patients requiring surgical re-intervention
Postoperative morbidity rate | Up to 30 days
  Postoperative surgical (bleeding, obstruction, postoperative ileus, abdominal collection, wound infection) and medical morbidity as well as mortality will be documented and graded according to the Dindo Clavien classification
Recovery times | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  Length of post-operative hospital stay, time to first flatus, time to first defecation, time to tolerance of liquid and solid diet will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Bucci, Prof, Principal Investigator — Federico II University of Naples
Locations (1):
- UOC Colonproctologia Chirurgica - Dipartimento di Medicina Clinica e Chirurgia - Università degli Studi di Napoli Federico II, Napoli, Italy

REFERENCES:
- [Background] Kono T, Ashida T, Ebisawa Y, Chisato N, Okamoto K, Katsuno H, Maeda K, Fujiya M, Kohgo Y, Furukawa H. A new antimesenteric functional end-to-end handsewn anastomosis: surgical prevention of anastomotic recurrence in Crohn's disease. Dis Colon Rectum. 2011 May;54(5):586-92. doi: 10.1007/DCR.0b013e318208b90f. PMID 21471760
- [Derived] Luglio G, Rispo A, Imperatore N, Giglio MC, Amendola A, Tropeano FP, Peltrini R, Castiglione F, De Palma GD, Bucci L. Surgical Prevention of Anastomotic Recurrence by Excluding Mesentery in Crohn's Disease: The SuPREMe-CD Study - A Randomized Clinical Trial. Ann Surg. 2020 Aug;272(2):210-217. doi: 10.1097/SLA.0000000000003821. PMID 32675483